CLINICAL TRIAL: NCT02909491
Title: Ionized Calcium and Behavioural Disorders in Older Adults (CALICO Study)
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016-36
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2016-09

CONDITIONS: Geriatric Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cases: Inpatient with severe behavioural disorders
- Controls: Inpatients without severe behavioural disorder and taking no antipsychotics

SUMMARY:
The primary objective of this study is to determine whether geriatric inpatients with severe behavioral disorders exhibit higher serum ionized calcium concentration than geriatric inpatients without behavioral disorders, but no difference in serum calcium or corrected calcium concentrations. The secondary objective of this study is to determine whether the serum ionized calcium concentration is associated with behavioral and cognitive performance among geriatric inpatients.

DETAILED DESCRIPTION:
Growing attention is paid to the neurological effects of calcium. While calcium is necessary for neuronal physiology, it appears that high serum calcium concentrations may be toxic to neurons. An analysis of the Rotterdam Study showed that, among older adults, higher concentrations of calcium were associated with greater cognitive disorders and faster cognitive decline. Similarly, delirium and behavioural disorders are reported in older adults with hypercalcemia. In contrast, other studies failed to find any association. For example, in France, an analysis of the EPIDOS study found no association between calcium concentration and cognitive performance. Thus, further studies remain necessary to make firmer conclusions about this link. In particular, it is interesting to note that all previous studies have used the serum concentrations of calcium or corrected calcium, but not yet ionized calcium. This assay is yet more reproducible, more sensitive and more correlated with clinical events. We propose that the non-use of ionized calcium assay may explain, at least in part, the discrepancies between previous studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 75 years and over
* Cases :

  * Inpatient with severe behavioural disorders
  * Being hospitalized in the geriatric acute care unit of Angers University Hospital, France
* Controls :

  * Inpatients without severe behavioural disorder and taking no antipsychotics
  * Being hospitalized in the geriatric acute care unit of Angers University Hospital, France
  * Paired on age (± 3 years) and gender

Exclusion Criteria:

* Inability to understand and speak French
* Opposition to the use of information collected for this research

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients are recruited in geriatric acute care.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-06; Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Comparison of serum ionized calcium concentrations between cases and paired controls. | This outcome is assessed at baseline.
  This measurement is assessed by a blood test.

SECONDARY OUTCOMES:
Comparison of serum corrected calcium concentration between cases and paired controls. | This outcome is assessed at baseline.
  This measurement is assessed by a blood test.
Comparison of the severity of behavioural disorders between cases and paired controls. | This outcome is assessed at baseline.
  The severity of behavioural disorders is assessed by a standardized scale (Frontotemporal Behavioural Rating Scale (FBRS), Lebert F. et Pasquier F., 1998)
Comparison of cognitive performance between cases and paired controls. | This outcome is assessed at baseline.
  Cognitive performance is assessed by the Mini-Mental State Examination (MMSE) score.

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: No